CLINICAL TRIAL: NCT03598738
Title: The Effect of Esomeprazole on Gastrin Levels and Glycaemic Regulation of Type 2 Diabetes: A Prospective Trial
Brief Title: The Effect of Esomeprazole on Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Yusuf Bozkuş, Assistant Professor, Baskent University Ankara Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA12/242
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Esomeprazole; Gastrin; HbA1c; Glycaemic Regulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Esomeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esomeprazole 40mg Group (Active Comparator): Intervention group consisted of 16 diabetic subjects that had various degrees of symptoms for functional dyspepsia, gastro-oesophageal reflux, gastritis or duodenitis. All of them were prescribed 40 mg of esomeprazole treatment for three months.
  Interventions: Drug: Esomeprazole 40mg
- Control Group (No Intervention): The control group consisted of without gastric complaints, thus who did not receive PPI drugs. This group was followed-up without any intervention for three months.

INTERVENTIONS:
Drug: Esomeprazole 40mg — Esomeprazole 40mg oral tablet, once a day
  Other Names: Nexium 40 mg
  Arms: Esomeprazole 40mg Group

SUMMARY:
The investigators aimed to prospectively investigate the effects of esomeprazole on glycaemic control in patients with type 2 diabetes mellitus. The investigators also aimed to associate this effect with gastrin levels. Thirty-two type 2 diabetes mellitus objects were recruited into intervention (n=16) and control (n=16) groups. The participants in the intervention group were prescribed 40 mg of esomeprazole treatment for three months. At the beginning of the study and at month 3, HbA1c level (%) and gastrin levels (pmol/L) of participants were assessed. Then the baseline and 3rd month data of groups were compared.

DETAILED DESCRIPTION:
Thirty-two patients recruited in the study. All the participants had a diagnosis of T2DM and had at least 1-year follow-up in Endocrinology outpatient clinic. All the study participants were chosen from regulated diabetic subjects whose diabetes treatment were not amended. The investigators excluded any cases needing revision in their treatment strategies due to ethical issues. Participants were recruited in intervention and control groups. Each group consisted of 16 diabetic subjects. Groups were matched for age, diabetes duration, body mass index, baseline HbA1c level and gastrin levels. In the intervention group, all participants had various degrees of symptoms for functional dyspepsia, gastro-oesophageal reflux, gastritis or duodenitis and all of them were prescribed 40 mg of esomeprazole treatment for three months. The control group consisted of without gastric complaints, thus who did not receive PPI drugs. This group was followed-up without any intervention for three months. All subjects were advised for dietary recommendations and lifestyle modifications. At the end of the study, all of them reported their adherence to these recommendations. Subjects, on pioglitazone and incretin-based therapies; subjects with a history of gastrointestinal surgery, liver or kidney disease, diabetic macro- or microvascular complications; who are lactating or pregnant, were excluded. Subjects on any PPI treatment or had a history of PPI use in a 3 months period before the study were not eligible.

The height was measured in the standing position with a tape measure fixed on the wall. Body weight, fat mass, and fat percentage were measured using a conventional bioelectrical impedance (BIA) device (TBF-300, Tanita corp., Tokyo, Japan). All measurements were completed after a mean period of 60 seconds. Subjects were asked not to consume alcohol during the 24-hour period before assessment and caffeine for the 4 hours before assessment. All accessories, such as heavy clothing, rings, and earrings, which could affect the measurements, were removed before the assessment. Body mass index was calculated as weight in kilograms divided by the square of the height in meters (kg/m2). All measurements were performed by one physician after the participants had fasted for at least 8 hours. Fasting blood glucose (FBG) (mg/dl.), triglyceride (mg/dL), high-density lipoprotein cholesterol (HDL-c, mg/dL), low-density lipoprotein cholesterol (LDL-c, mg/dL), thyroid-stimulating hormone (TSH) (IU/mL), HbA1c level (%) and gastrin levels (pmol/L) were measured by using a sample of venous blood. TSH assays were performed via immunochemiluminescent assay (Architect c8200, Abbott). FBG, LDL-c, HDL-c, and triglyceride levels were measured by using the hexokinase 7/G-6-PDH method, a measured liquid-selective detergent method, an accelerator-selective detergent method, and a glycerol phosphate oxidase method (Architect c8200, Abbott), respectively. HbA1c was via the enzymatic method using Architect c4000 (Abbott) system from human complete blood and hemolysate. Serum gastrin level was measured by a competitive radioimmunoassay using a rabbit antiserum raised against a gastrin 17 albumin conjugate (DiaSource ImmunoAssasys S.A., Louvain-la-Neuve, Belgium). According to the manufacturer, the range of gastrin level is 11-54 pmol/L and the lowest detectable concentration is 5 pmol/L. All measurements were performed both at baseline and the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* All the participants that has a diagnosis of T2DM and had at least 1-year follow-up in Endocrinology outpatient clinic.
* All the study participants were chosen from regulated diabetic subjects whose diabetes treatment were not amended.
* In the intervention group, all participants had various degrees of symptoms for functional dyspepsia, gastro-oesophageal reflux, gastritis or duodenitis
* The control group consisted of without gastric complaints, thus who did not receive PPI drugs.

Exclusion Criteria:

* We excluded any cases needing revision in their treatment strategies due to ethical issues.
* Subjects, on pioglitazone and incretin-based therapies;
* Subjects with a history of gastrointestinal surgery, liver or kidney disease, diabetic macro- or microvascular complications;
* Subjects who are lactating or pregnant
* Subjects on any PPI treatment or had a history of PPI use in a 3 months period before the study, were excluded.

Ages: 47 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
HbA1c change | 3 months
  HbA1c change with esomeprazole in 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Bozkuş, Assist Prof, Study Director — Başkent University Endocrinolgy Dep; Neslihan Başçıl Tütüncü, Prof, Principal Investigator — Başkent University Endocrinolgy Dep; Özlem Turhan İyidir, Assoc Prof, Principal Investigator — Başkent University Endocrinolgy Dep; Umut Mousa, Dr, Principal Investigator — Başkent University Endocrinolgy Dep; Nazlı Kırnap, Dr, Principal Investigator — Başkent University Endocrinolgy Dep; Canan Çiçek Demir, Dr, Principal Investigator — Başkent University Endocrinolgy Dep; Aslı Nar, Assoc Prof, Principal Investigator — Başkent University Endocrinolgy Dep

IPD SHARING:
Plan to Share IPD: Undecided